CLINICAL TRIAL: NCT05948163
Title: Caries Risk Assessment Using ADA Tool Among A Group of Egyptian Children in Mixed Dentition Stage : A Cross-Sectional Study
Brief Title: Caries Risk Assessment in Egyptian Children in Mixed Dentition Stage
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Yehia Zekry Ibrahim, Doctor, Cairo University
Other Study IDs: ADA tool
Record Dates: First submitted 2023-07-08; First posted 2023-07-17 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Caries Risk Assesment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aim to assess the validity of ADA caries risk assessment tool on the Egyptian Children in mixed dentition stage .

DETAILED DESCRIPTION:
Dental caries is the most common chronic disease of childhood that causes health problems such as pain and infection in children reducing their quality of life.

Risk for caries includes physical, biological, environmental, behavioral, and lifestyle-related factors as insufficient fluoride exposure, poor oral hygiene,inappropriate methods of feeding infants, and poorness .

Risk is a probability that an event will occur. Caries Risk Assessment (CRA) is "prediction of future caries based on the diagnosis of current disease by evaluation of risk and protective factors for making evidence-based clinical decisions. Individual risk assessment constitutes the cornerstone of the treatment plan for the management of early childhood caries for pediatric patients. Caries risk assessment should be included in the treatment plan to facilitate The decision-making process concerning preventive care (both home and office) treatment, recall appointments.

An ideal risk assessment model should be inexpensive, easy to use and time efficient with a high degree of accuracy in caries predictive value.

American Dental Association (ADA) is a tool for caries risk assessment and Management , that when modified to meet the needs of an environment Will be of tremendous use in caries risk assessment. The ADA's mission is to help dentists succeed and support the advancement of the health of the public.

ELIGIBILITY:
Inclusion Criteria:

* Children age range from 6 to 12 years.
* Apparently healthy children.
* Children affected by dental caries.
* Parents acceptance for their children's participation in the study.

Exclusion Criteria:

* Children on long-term medication.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 6 to 12 years
Sampling Method: Non-Probability Sample
Enrollment: 296 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Caries Risk Assessment using ADA | one year
  Measurement Method Questions Measurement Method :Questions